CLINICAL TRIAL: NCT01959269
Title: RECORA- Regorafenib in Patients With Metastatic Colorectal Cancer (mCRC) After Failure of Standard Therapy.
Brief Title: Investigating the Use of Regorafenib (Stivarga®) in Patients With Metastatic Colorectal Cancer (mCRC) After Failure of Standard Therapy
Acronym: RECORA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16665; SV1313 (Other: Company internal)
Record Dates: First submitted 2013-10-08; First posted 2013-10-09 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Regorafenib: Patients treated with Stivarga as 3rd or 4th line treatment, no intervention
  Interventions: Drug: Regorafenib (Stivarga, BAY 73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY 73-4506) — As determined by the treating physician

SUMMARY:
The purpose of the study is to investigate the safety and effectiveness of Stivarga in patients with metastatic colorectal carcinoma in routine use in Germany. The study is purely observational, only data from routine treatment are to be collected. The treatment and treatment conditions are solely at discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:´

* Male or female patients ≥ 18 years of age with metastatic CRC for whom the decision has been taken by the investigator to treat with Stivarga.
* Patients must have signed an informed consent form

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients ≥ 18 years of age with a diagnosis of metastatic colorectal carcinoma (mCRC) will be enrolled in the sites during the enrollment period. All treatment decisions prior inclusion of a patient as well as during the observation must be made by the investigator based on his regular medical practice. Patients must give written informed consent prior to documentation.
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | after 40 months

SECONDARY OUTCOMES:
Progression-free survival | after 40 months
Time to progression | after 40 months
Disease control rate (DCR) | after 40 months
  Disease control rate (DCR) is defined as percentage of patients, whose best response was not progressive disease (i.e. complete response, partial response or stable disease).
Duration of Stivarga treatment | after 40 months
  Duration of Stivarga treatment is defined as the time interval from start of Stivarga therapy to the date of permanent discontinuation of Stivarga therapy (regardless of the reason for discontinuation)
Tumor status at different visits | after 40 months
  The tumor status at different visits will be evaluated according to the categories "complete response", "partial response", "stable disease", "progressive disease by clinical judgment", "progressive disease measurement proven", "unknown" and "not applicable". The best overall response will be analyzed providing absolute and relative frequencies of the tumor status categories.
Incidence of treatment emergent adverse events (TEAE) | after 18 and 40 months
  Detailed information collected for each TEAE will include: a description of the event, duration, whether the TEAE was serious, relationship to Stivarga, action taken, clinical outcome. Summary tables will present the number of subjects observed with TEAEs and corresponding percentages. Additional subcategories will be based on event intensity and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Germany